CLINICAL TRIAL: NCT02645903
Title: Ultrasound-guided Transversus Abdominis Plane Block for Postoperative Analgesia in Living Donor Hepatectomy: Randomized Controlled Double-blinded Trial
Brief Title: Transversus Abdominis Plane Block for Postoperative Analgesia in Living Donor Hepatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Erdoğan, Associted professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAP
Record Dates: First submitted 2015-12-24; First posted 2016-01-05 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Acute Pain
Keywords: transversus abdominis plane block; living liver transplantation; postoperative analgesia
MeSH Terms: conditions — Acute Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transversus abdominis plane block (Active Comparator): Patients who received a tranversus abdominis plane block with ultrasound after standard general anesthesia represented Group 1.
  The tranversus abdominis plane block was performed bilaterally by obtaining an image with real time ultrasound guidance with a 6-13 MHz linear probe.
  The block was placed with a 22 G 80 mm needle while obtaining real-time images via an in-plane technique.
  Two 20 mL syringes were prepared after preparing a local anesthetic concentration of 1.5 mg/kg of 0.5% bupivacaine to 40 mL with saline. These were administered to the left and right abdominal walls.
  Postoperative analgesia was administered through a morphine the patient-controlled analgesia device.
  Interventions: Drug: Transversus Abdominis Plane Block
- nonblocked (Placebo Comparator): Patients who received standard general anesthesia alone made up Group 2. Postoperative analgesia was administered through a morphine the patient-controlled analgesia device.
  Interventions: Drug: standard general anesthesia

INTERVENTIONS:
Drug: Transversus Abdominis Plane Block — Cases to whom used bupivacaine with ultrasound guided transversus abdominis plane block was applied after standard general anesthesia were determined as Group 1
  Other Names: Marcaine plain+morphine
  Arms: transversus abdominis plane block
Drug: standard general anesthesia — Cases to whom applied alone standard general anesthesia were determined as Group 2
  Other Names: morphine
  Arms: nonblocked

SUMMARY:
Living donor organ transplantation has increased in recent years due to an increased need for organs. The objective of this study was to investigate the effects of a TAP block on postoperative analgesia and opioid consumption in liver transplantation donors in whom a right lateral extending upper mid-line abdominal incision was used.

DETAILED DESCRIPTION:
This prospective randomized controlled double-blinded study was conducted with 50 liver transplantation donors between 18-65 years who were scheduled to undergo right hepatectomy surgery. Cases to whom TAP block with ultrasound was applied after standard general anesthesia were determined as Group 1 and cases to whom only standard general anesthesia was applied, were determined as Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplantation donors

Exclusion Criteria:

* Patients with a history of allergy to the drugs used in the study protocol, coagulation pathology, opioid tolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
pain scores (at movement and at rest) | postoperatively at 24 hours
  Pain scores were assessed using a visual analog scale (0: No pain, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10: Excruciating pain).

SECONDARY OUTCOMES:
morphine consumption | postoperatively at 24 hours
  morphine consumption were measured in postoperatively 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ali Erdogan, Principal Investigator — Inonu University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdallah FW, Chan VW, Brull R. Transversus abdominis plane block: a systematic review. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):193-209. doi: 10.1097/AAP.0b013e3182429531. PMID 22286518